CLINICAL TRIAL: NCT01888835
Title: Mirtazapine for the Treatment of Methamphetamine Dependence Among MSM: a 6-month Randomized Controlled Trial With 3 Months of Follow-up
Brief Title: Mirtazapine for the Treatment of Methamphetamine Dependence Among MSM (M2.0)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Phillip Coffin, MD, MIA (Other Government)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Phillip Coffin, MD, MIA, Director, Substance Use Research Unit, San Francisco Department of Public Health
Organization: San Francisco Department of Public Health (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1R01DA034527 (NIH); R01DA034527 (NIH)
Record Dates: First submitted 2013-06-25; First posted 2013-06-28 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Amphetamine-Related Disorders
Keywords: HIV; sexual behavior
MeSH Terms: conditions — Amphetamine-Related Disorders; Sexual Behavior | interventions — Mirtazapine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mirtazapine (Active Comparator): mirtazapine 30 mg orally per day
  Interventions: Drug: Mirtazapine
- Placebo (Placebo Comparator): placebo (30 mg) orally per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mirtazapine
  Other Names: Remeron
  Arms: Mirtazapine
Drug: Placebo
  Arms: Placebo

SUMMARY:
The investigators recently conducted a double-blind, randomized controlled trial (n=60) of limited duration (12 weeks), and found that compared with placebo, oral mirtazapine, an FDA-approved antidepressant, significantly reduced meth use in those receiving mirtazapine, as determined by reduction in meth-positive urines. Sexual risk behaviors also declined significantly in the mirtazapine arm compared to placebo. Mirtazapine decreased meth use despite low adherence: by medical event monitoring system (MEMS) caps, only 48.5% of daily doses were taken. All participants received weekly substance use counseling and monthly, brief clinician-delivered adherence counseling. The investigators propose expanding upon these results by lengthening the treatment period to 24 weeks, with adherence reminders added to the counseling, and determining if efficacy is sustained up to 12 weeks after drug discontinuation. The sample size for this 9-month study is 120.

ELIGIBILITY:
Inclusion Criteria:

1. born male, or born female and does not identify as female;
2. reports anal sex with men in the prior three months while under the influence of meth;
3. diagnosed with meth dependence by SCID;
4. interested in stopping or reducing meth use;
5. at least one meth-positive urine during screening and run-in period;
6. no current acute illness requiring prolonged medical care;
7. no serious chronic illnesses that are likely to progress clinically during trial participation;
8. able and willing to provide informed consent and adhere to visit schedule;
9. age 18-69 years;
10. baseline CBC, total protein, albumin, glucose, alkaline phosphatase, creatinine, BUN, and electrolytes without clinically significant abnormalities as determined by clinician in conjunction with symptoms, physical exam, and medical history
11. current CD4 count ≥ 200 cells/mm3; or CD4 count of 100 - 199 cells/mm3 and HIV viral load < 200 copies/mL
12. text-capable cell phone or access to email

Exclusion Criteria:

1. Evidence of current major depression by SCID;
2. history of bipolar disorder or psychotic disorder, as determined by SCID;
3. known allergy or previous adverse reaction to mirtazapine;
4. taking an anti-depressant medication within the past 30 days, including mirtazapine or a monoamineoxidase inhibitor;
5. moderate or severe liver disease (AST, ALT, and total bilirubin >= 5 times upper limit of normal);
6. impaired renal function (estimated GFR <40 ml/min);
7. currently participating in another research study;
8. pending legal proceedings with high risk for incarceration during the time of planned study participation;
9. any condition that, in the principal investigator's judgment, interferes with safe study participation or adherence to study procedures.

Ages: 18 Years to 69 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-08; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Number of methamphetamine-positive urine tests | weekly for 9 months
  To determine the efficacy of mirtazapine vs placebo at 12 weeks and 24 weeks of treatment plus counseling, and to determine whether efficacy is sustained for an additional 12 weeks after discontinuation of treatment and counseling (weeks 24 to 36).

SECONDARY OUTCOMES:
Sexual risk (see description) | 9 months
  To assess if the intervention reduces HIV risk behaviors, including number of male sex partners, number of male anal sex partners with whom meth is used and episodes of unprotected anal sex with serodiscordant partners.

OTHER OUTCOMES:
Adherence to study drug | 6 months
  To measure the acceptability of mirtazapine and placebo by determining (via electronic pill boxes and self-report) medication adherence including percent of doses taken, taking less than 80% of medication, patterns of non-adherence (e.g. use every other day, during the weekend, longer alternating periods on and off medication), and time to stopping medication.
Number of adverse events | 6 months
  To measure the tolerability of mirtazapine and placebo, as determined by the number of adverse clinical events in the mirtazapine and placebo arms.

CONTACTS AND LOCATIONS:
Overall Officials: Phillip O Coffin, M.D., Principal Investigator — San Francisco Department of Public Health; Steven L Batki, M.D., Principal Investigator — University of California, San Francisco; Emily Behar, Study Director — San Francisco Department of Public Health
Locations (1):
- Substance Use Research Unit, San Francisco, California, United States

REFERENCES:
- [Derived] Coffin PO, Santos GM, Hern J, Vittinghoff E, Walker JE, Matheson T, Santos D, Colfax G, Batki SL. Effects of Mirtazapine for Methamphetamine Use Disorder Among Cisgender Men and Transgender Women Who Have Sex With Men: A Placebo-Controlled Randomized Clinical Trial. JAMA Psychiatry. 2020 Mar 1;77(3):246-255. doi: 10.1001/jamapsychiatry.2019.3655. PMID 31825466